CLINICAL TRIAL: NCT00714948
Title: Phase II Study of Gemcitabine and Split-dose Cisplatin (GC) Plus Sorafenib in Chemotherapy-naïve Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: Gemcitabine and Split-dose Cisplatin (GC) Plus Sorafenib in Chemotherapy-naïve Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-168
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-10

CONDITIONS: Bladder Cancer; URINARY BLADDER
Keywords: Bladder; Urinary; SORAFENIB; CISPLATIN; GEMCITABINE
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin; Sorafenib

ARMS (1):
- 1 (Experimental): This is a phase II trial of gemcitabine and Split-dose cisplatin plus sorafenib.
  Interventions: Drug: gemcitabine and cisplatin plus sorafenib

INTERVENTIONS:
Drug: gemcitabine and cisplatin plus sorafenib — Gemcitabine 1000 mg/m 2 will be administered on days 1 and 8 and cisplatin 35 mg/m 2 will be administered on days 1 and 8. A total of six cycles of therapy will be administered at 21day intervals. Sorafenib 400 mg PO twice daily will be initiated on day 1 of cycle 1 and continued, as tolerated, until the time of disease progression or a maximum of 12 months. The total chemotherapy dose for gemcitabine and cisplatin (GC) may be modified for patients with severe obesity (e.g. body surface area (BSA) > 2.1), after consultation with the Principal Investigator.

SUMMARY:
Standard chemotherapy drugs generally work by killing rapidly dividing cells in your body. Cancers cells are some of the most rapidly dividing cells and that is why chemotherapy can be effective in some patients. Gemcitabine and Cisplatin are an effective and standard drug combination used to treat locally advanced and metastatic urothelial cancer. However, these drugs do not shrink tumors in all patients and when they do, it is generally for a limited amount of time. This has led scientists to look for different ways to treat cancer.

New drugs have been developed to treat cancer that work differently than standard chemotherapy drugs. These drugs attempt to decrease the blood supply to tumors. By doing so, this may limit the tumor's source of oxygen and nutrients and prevent the tumor from growing. Sorafenib is an example of a drug that works in this way.

In some patients with advanced kidney cancer, sorafenib alone has been shown to slow the progression of their disease. The purpose of this study is to find out what effects, good and/or bad, the combination of gemcitabine, cisplatin, and sorafenib has on you and your cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable or evaluable urothelial cancer.

  * Measurable disease includes unresectable or metastatic urothelial tract tumors that are unidimensionally measurable by xray,CT/MRI scan or physical examination.
  * Evaluable disease is restricted to patients with unresectable primary bladder tumors which can be evaluated for response by cystoscopy.
* Pathologic confirmation by the Department of Pathology at MSKCC.
* Karnofsky Performance Status (KPS) ≥60%.
* Adequate marrow function defined as granulocytes ≥ 1500 cells/mm 3 , platelets ≥ 100,000 cells/mm 3 , and hemoglobin ≥ 8.0 g/dl.
* Serum creatinine < 2.0 mg/dl
* 24-hour urine sample demonstrating creatinine clearance ≥ 60 ml/min/1.73m2 or calculated creatinine clearance ≥ 60 ml/min/1.73m 2 using the formula: Jeliffe Equation: estimated creatinine clearance = 98 x (0.8 [age(yrs) 20]/Serum Creatinine (mg/dL) x (0.9 if Female))
* Adequate hepatic function defined as:

  * Total Bilirubin < or = to 1.5 x ULN
  * AST and ALT < or = to 3.0 x ULN (< or = to 5.0 x ULN is acceptable if liver has tumor involvement)
* Normal coagulation profile including PT/INR and PTT, unless patient is receiving anticoagulation therapy with agents such as warfarin or heparin.
* Age ≥ 18 years
* Informed consent
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Patients are encouraged to continue barrier method contraception for two years or longer after treatment.

Exclusion Criteria:

* Prior treatment with systemic chemotherapy (prior intravesical therapy is permitted).
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.
* Blood Pressure of > 150/100 mm Hg.
* Irradiation within 4 weeks of start of protocol.
* Evidence of another active cancer, except for nonmelanoma skin carcinoma, insitu carcinoma of the cervix curatively treated, and adenocarcinoma of the prostate that has been surgically treated with a post-treatment PSA that is nondetectable.
* Significant cardiovascular disease including congestive heart failure (New York Heart Association Class II or higher) or active angina pectoris.
* History of a myocardial infarction within 6 months.
* History of a stroke or transient ischemic attack within 6 months.
* Clinically significant peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* Presence of central nervous system or brain metastases.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0.
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0.
* History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to Day 0.
* Serious nonhealing wound, ulcer, or bone fracture.
* History of persistent gross hematuria.
* Uncontrolled infection.
* Hypersensitivity to sorafenib, or any component of the formulation.
* Pregnant (positive pregnancy test) or lactating.
* Inability to comply with the study and/or followup procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Milowsky, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: 07/10/2008 Protocol Closed to Accrual:12/08/2009 Primary Completion Date: 11/22/2011 Recruitment Location is the medical clinic
Groups:
- Gemcitabine and Split-dose Cisplatin + Sorafenib: This is a phase II trial of gemcitabine and Split-dose cisplatin plus sorafenib.
  Gemcitabine 1000 mg/m 2 will be administered on days 1 and 8 and cisplatin 35 mg/m 2 will be administered on days 1 and 8. A total of six cycles of therapy will be administered at 21day intervals. Sorafenib 400 mg PO twice daily will be initiated on day 1 of cycle 1 and continued, as tolerated, until the time of disease progression or a maximum of 12 months.
Period: Overall Study
Arm/Group | Gemcitabine and Split-dose Cisplatin + Sorafenib
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine and Split-dose Cisplatin + Sorafenib
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Progression Free Survival Rate at One Year Untreated Patients With Advanced/Metastatic Urothelial Carcinoma Treated With the Combination of Sorafenib, Gemcitabine, and Cisplatin.
Time Frame: conclusion of the study
Arm/Group | Gemcitabine and Split-dose Cisplatin + Sorafenib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Gemcitabine and Split-dose Cisplatin + Sorafenib
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Split-dose Cisplatin + Sorafenib (N=2)
Bladder infection (Infections and infestations) | 1 (1)
Thromboembolic event (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Split-dose Cisplatin + Sorafenib (N=2)
Alanine aminotransferase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (10)
Creatinine increased (Investigations) | 2 (15)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Edema: limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (31)
Anemia (Blood and lymphatic system disorders) | 2 (23)
Hemorrhage, Urinary NOS (Renal and urinary disorders) | 1 (2)
INR increased (Investigations) | 1 (5)
White blood cell decreased (Investigations) | 2 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (11)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (7)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3)
Platelet count decreased (Investigations) | 2 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (7)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (8)
Urinary frequency (Renal and urinary disorders) | 1 (5)
Vomiting (Gastrointestinal disorders) | 2 (3)
Weight loss (Investigations) | 2 (6)

LIMITATIONS AND CAVEATS:
Early termination leading to no subjects analyzed. Only two participants were enrolled and treated on this study. Neither completed the study as they both came off due to adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes